CLINICAL TRIAL: NCT06183021
Title: The Effect of Cryotherapy on the Outcome of Pulpotomy and Root Canal Treatment of Deep Dentinal Caries: a Randomized Clinical Trial.
Brief Title: The Effect of Cryotherapy on the Outcome of Pulpotomy and Root Canal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cangül Keskin, Associate professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5502
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Pulpitis; Caries; Dentin; Pain, Postoperative
Keywords: vital pulp treatment; cryotherapy; quality of life
MeSH Terms: conditions — Pulpitis; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Total pulpotomy with cryotherapy (Experimental): Total coronal amputation will be performed using vital pulp cryotherapy
  Interventions: Procedure: Vital pulp cryotherapy
- Total pulpotomy (No Intervention): Total coronal amputation will be performed.
- Root canal treatment with cryotherapy (Experimental): Orthograde root canal treatment will be performed with intracanal cryotherapy.
  Interventions: Procedure: Intracanal cryotherapy
- Root canal treatment (No Intervention): Orthograde root canal treatment will be performed.

INTERVENTIONS:
Procedure: Vital pulp cryotherapy — Shaved ice made from sterile distilled water will be applied around the treated tooth especially in contact with amputated pulp tissue until totally dissolves.
  Arms: Total pulpotomy with cryotherapy
Procedure: Intracanal cryotherapy — After mechanical preparation, a 5-minute final irrigation with 20 mL cold saline (2.5 Centigrade degrees) will be applied using a negative pressure irrigation technique per canal.
  Arms: Root canal treatment with cryotherapy

SUMMARY:
The goal of this randomized clinical trial is to compare the outcome of total amputation and root canal treatment with or without cryotherapy in terms of postoperative pain, quality of life, and treatment success for the management of deep dentinal caries. The main questions it aims to answer are:

Does cryotherapy influence the outcome, life quality and treatment success in total pulpotomy? Does cryotherapy influence the outcome, life quality and treatment success in root canal treatment? Does the outcome of total pulpotomy and root canal treatment differ in cases of pulpitis?

There are 4 experimental groups:

1. Total pulpotomy with cryotherapy group
2. Total pulpotomy group (Control 1)
3. Root canal treatment with cryotherapy group
4. Root canal treatment group (Control 2)

DETAILED DESCRIPTION:
Sample Size Determination Method and Total Number of Subjects for the Study:

The study will span 24 months, and a total of 144 patients meeting the inclusion criteria will be selected from those seeking treatment at the Endodontics clinic of Ondokuz Mayıs University Faculty of Dentistry.

An a priori power analysis was performed using the treatment success rate parameter under the "Survival Analysis: Comparison of Two Survival Curves - Lachin" section at the link: Survival Analysis: Comparison of Two Survival Curves - Lachin. Based on the treatment success rates in the study by Asgary et al. (2015) - 76.1% for vital pulp therapy and 75.6% for root canal treatment, with a type I error of 0.05 and a beta value of 0.95, a minimum sample size of 30 per group was calculated. Considering a 20% follow-up loss, 36 subjects per group will be included (n = 36).

Patients within the age range of 18-65, systemically healthy, with upper and lower jaw molars, deep dentin caries, and no known allergies to materials and drugs used in root canal treatment, will be assessed for inclusion criteria in the endodontics clinic. Pulp sensitivity tests using cold and electric pulp tests will be conducted. If the pulp chamber does not become exposed after caries removal or if necrosis is detected in at least one canal (with no bleeding) after cavity preparation, the voluntary participant will be excluded from the study, and appropriate treatment will be completed. Radiological examination will evaluate the presence of radiolucent lesions in periapical areas using periapical radiographs taken from different angles. Teeth with a periapical index value greater than 1, indicating radiolucency observed in apical periodontitis, will be excluded (Orstavik 1986). Teeth that cannot be isolated with a rubber dam, for which coronal obturation cannot be achieved, teeth with fractures, advanced periodontal disease, and teeth with multiple lost cavity walls will be excluded from the study.

Before starting the treatment, patients will randomly select one of four sealed envelopes containing the name of the study group. The envelope will be sealed until the randomization phase (before cavity preparation after local anaesthesia and isolation) to ensure that the operator remains unaware of the study group name. Patients will be informed about the visual analogue scale (VAS) and quality of life scales related to oral health before the treatment.

Preparation and Disinfection for Treatment:

The tooth will be isolated with a rubber dam after local anaesthesia administration (2.0 mL adrenaline 1:100,000 4% articaine). Following isolation, the coronal surfaces of the tooth will be sequentially disinfected with 3% hydrogen peroxide and 5.25% sodium hypochlorite. The investigator will perform all operative procedures under 3.5x magnification using loupes available in our clinic.

Number and Names of Groups in the Study:

Total Coronal Amputation Cryotherapy and Control Groups:

In this group, the coronal pulp exposed after caries removal will be completely removed with a sterile steel round bur. In the cryotherapy subgroup, the cavity surface will be treated with 1 minute of grated sterile ice, applied according to the protocol described by Bahcall et al. (2019), and removed with a melting water absorbent. The pulp chamber will be irrigated in both groups with 17% ethylenediaminetetraacetic acid (EDTA) for 1 minute. Subsequently, the pulp chamber will be restored with a composite resin over a Biodentine-prepared cavity using light-cured composite resin. If bleeding persists for more than 5 minutes in the pulp chamber, the participant will be excluded, and root canal treatment will be completed.

Root Canal Treatment Cryotherapy and Control Groups:

After cleaning the caries, an appropriate endodontic access cavity will be prepared. Using a size 10-15 K-type hand file with an apex locator, canal shaping will be performed with the TruNatomy file system. After each change, preserving apical patency will be ensured with a size 10-15 K-type file. After preparation, the canals will be irrigated sequentially with 5 mL of 17% EDTA, distilled water, and 5.25% sodium hypochlorite.

In the control group, the EndoVac negative-pressure irrigation system will be used to irrigate with 20 mL of distilled water stored at room temperature for 5 minutes. In the cryotherapy group, the same irrigation system will be used to irrigate with 20 mL of distilled water stored at 2.5°C in the refrigerator for 5 minutes. Temperature control will be ensured during irrigation using thermocouples and a thermometer. The canals will then be dried with sterile paper points and filled with AH Plus Bioceramic and gutta-percha points. Coronal restorations will be performed with light-cured composite resin and bond adhesive.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-65.
* Having an upper or lower jaw molar with deep dentin caries.
* No previous restorations, root canal treatments, fractures, or cracks in the relevant tooth.
* Loss of substance in the relevant tooth is limited to a Class I type, involving only the occlusal surface of the tooth.
* Obtaining a negative response to palpation and percussion.
* Normal periodontal tissues (pocket depth less than 3 mm and normal mobility).
* Exposing the pulp when the caries is completely cleaned

Exclusion Criteria:

* Having a chronic systemic disease that impedes local anaesthesia and the application of endodontic procedures.
* Presence of cracks, fractures, or restorations in the relevant tooth.
* Raynaud's phenomenon.
* Partial or total necrosis in the relevant tooth.
* Teeth with cavities other than Class I, involving more than one surface of substance loss in the relevant tooth.
* Teeth diagnosed with acute apical abscess or chronic apical abscess.
* Pregnant or breastfeeding women.
* History of allergy to materials and drugs used in treatment.
* Patients reporting spontaneous pain with a Visual Analog Scale (VAS) score of 5 or above and provoked pain lasting over 20 seconds during examination.
* Positive response to percussion and palpation.
* Advanced periodontal disease (Pocket depth greater than 3 mm and Class I or higher mobility).
* Pulp not exposed when caries is cleaned (not emerging, covered with intact dentin).
* The root apex of the relevant tooth being immature

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessment | 1st day, 2nd day, 7th day after intervention
  Postoperative pain will be assessed using visual analogue scale with a 10 cm straight line with one end meaning no pain (0) and the other end meaning the worst pain imaginable (10) and anchor markings at each millimeter
Oral health related quality of life questionnaire consisted of 14 questions | 1st week, 6th month after intervention
  Oral health related quality of life scale will be applied
Treatment success based on clinical and radiographic examination | 1st week, 3rd month, 6th month
  The periapical health and tooth/pulp survival

CONTACTS AND LOCATIONS:
Overall Officials: Cangül Keskin, PhD, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University Dp. Endodontics, Faculty of Dentistry, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duncan HF, El-Karim I, Dummer PMH, Whitworth J, Nagendrababu V. Factors that influence the outcome of pulpotomy in permanent teeth. Int Endod J. 2023 Mar;56 Suppl 2:62-81. doi: 10.1111/iej.13866. Epub 2022 Nov 22. PMID 36334098
- [Background] Elmsmari F, Ruiz XF, Miro Q, Feijoo-Pato N, Duran-Sindreu F, Olivieri JG. Outcome of Partial Pulpotomy in Cariously Exposed Posterior Permanent Teeth: A Systematic Review and Meta-analysis. J Endod. 2019 Nov;45(11):1296-1306.e3. doi: 10.1016/j.joen.2019.07.005. Epub 2019 Sep 10. PMID 31515048
- [Background] Cushley S, Duncan HF, Lappin MJ, Tomson PL, Lundy FT, Cooper P, Clarke M, El Karim IA. Pulpotomy for mature carious teeth with symptoms of irreversible pulpitis: A systematic review. J Dent. 2019 Sep;88:103158. doi: 10.1016/j.jdent.2019.06.005. Epub 2019 Jun 20. PMID 31229496